CLINICAL TRIAL: NCT02736799
Title: Effect of Vibrant Capsule on Gastric Emptying and Antropyloroduodenal Motility in Healthy Volunteers: A Sham Device Controlled, Single Center Pilot Study
Brief Title: Effect of Vibrant Capsule on Gastric Emptying and Antropyloroduodenal Motility in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 215CLD
Record Dates: First submitted 2016-03-30; First posted 2016-04-13 (Estimated); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sham vibrating capsule (Sham Comparator): Sham vibrating capsule
  Interventions: Device: Sham vibrating capsule
- Vibrant Capsule (1 vibration) (Active Comparator): 1 vibration/min
  Interventions: Device: Vibrant Capsule (1 vibration)
- Vibrant Capsule (3 vibration) (Active Comparator): 3 vibrations/min
  Interventions: Device: Vibrant Capsule (3 vibration)
- Vibrant Capsule (5 vibration) (Active Comparator): 5 vibrations/min
  Interventions: Device: Vibrant Capsule (5 vibration)

INTERVENTIONS:
Device: Sham vibrating capsule — Sham device without vibration
  Arms: Sham vibrating capsule
Device: Vibrant Capsule (1 vibration) — 1 vibration/min
  Arms: Vibrant Capsule (1 vibration)
Device: Vibrant Capsule (3 vibration) — 3 vibration/min
  Arms: Vibrant Capsule (3 vibration)
Device: Vibrant Capsule (5 vibration) — 5 vibration/min
  Arms: Vibrant Capsule (5 vibration)

SUMMARY:
The Vibrant capsule is a novel vibrating device for the treatment of gastrointestinal disorders. The effect of different vibrations on the motor functions of the gastrointestinal tract are unclear. The study will focus on the stomach in healthy volunteers.

The study will compare the effects of Vibrant capsule treatment and Sham capsule treatment on gastric emptying and gastric motility in healthy volunteers.

DETAILED DESCRIPTION:
Healthy volunteers participants were randomized to one of 4 treatment groups: sham VIBRANT or vibrating VIBRANT capsule at rates of 1, 3 or 5 per minute. The studies were conducted in one day.

Following an overnight fast, participants underwent introduction of the multilumen manometric catheter into the proximal small intestine with sensors across the antroduodenal junction. A 4-meter Teflon® (green) guidewire and manometry tube were placed transnasally and advanced into the duodenum with the distal end of the manometry tube within the distal duodenum or proximal jejunum.

Following placement of the manometry tube a 30 minute baseline motility assessment was performed followed by the first of two VIBRANT OR SHAM VIBRANT CAPSULES administered as randomly assigned. Motility assessment performed for an additional 25-30 minutes before the digestion of the standardized breakfast test meal. A single spot image will be obtained to document the location of the capsule prior to the meal.

Approximately thirty minutes following ingestion of the capsule, participants ingested a standardized breakfast meal (320kcal egg, toast, milk) containing 99mTc. Anterior and posterior gamma camera images obtained immediately following ingestion of the meal and every 15 minutes until 240 minutes. In addition, every 30 minutes one hundred millimeter Visual analog scales (VAS) recorded to assess levels of nausea, fullness, gas, and abdominal pain.

Participants were seated in a semi-recumbent position (~45 degrees) for recording motility and obtaining anterior scintigraphy images simultaneously. Following the 90-minute scan, the participants ingested a second active VIBRANT or sham capsule. Subsequent scans continued at scheduled intervals until 240 minutes after the test meal ingestion to complete the assessment of gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent prior to any study procedures, and be willing and able to comply with study procedures
2. No medical problems or chronic diseases, specifically, no type 2 diabetes mellitus
3. Body mass index of 18-35 kg/m2
4. Female subjects must have negative urine pregnancy tests and must not be lactating prior to receiving study medication and radiation exposure. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. Female subjects unable to bear children must have this documented in the medical record [i.e., tubal ligation, hysterectomy, or post-menopausal (defined as a minimum of one year since the last menstrual period)].

Exclusion Criteria:

1. Unable or unwilling to provide informed consent or to comply with study procedures
2. Diagnosis of gastrointestinal diseases
3. Structural or metabolic diseases that affect the gastrointestinal system
4. Unable to avoid the following over-the-counter medications 48 hours prior to the baseline period and throughout the study:

   1. Medications that alter gastrointestinal transit including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin
   2. Analgesic drugs including Nonsteroidal Anti-Inflammatory Drugs and COX-2 inhibitors NOTE: stable doses of thyroid replacement, estrogen replacement, low-dose aspirin for cardioprotection, and birth control (but with adequate backup contraception as drug-interactions with birth control have not been conducted) are permissible.
5. History of recent surgery (within 60 days of screening)
6. Acute or chronic illness or history of illness which, in the opinion of the investigator, could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data, such as frequent angina, Class III or IV congestive heart failure, moderate impairment of renal or hepatic function, poorly controlled diabetes, etc.
7. Any clinically significant abnormalities on physical examination or laboratory abnormalities identified in the medical record, as determined by the investigator
8. Acute gastrointestinal illness within 48 hours of initiation of the baseline period
9. Females who are pregnant or breastfeeding
10. History of excessive alcohol use or substance abuse
11. Participation in an investigational study within the 30 days prior to dosing in the present study
12. Any other reason, which in the opinion of the investigator, would confound proper interpretation of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 1
Not completed — stopped study after receipt of Capsule #1 due to sore throat. | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (15.80) | 38.17 (18.05) | 28.5 (10.82) | 28.17 (10.26) | 32 (13.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 4 | 15
  Male | 3 | 2 | 2 | 2 | 9
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.75 (3.02) | 26.3 (4.97) | 26.83 (1.89) | 26.73 (4.745) | 26.57 (3.66)

OUTCOME MEASURES:

1. Primary Outcome: Gastroduodenal Manometry Measurement
Description: The main outcome measure is the Gastro-duodenal manometry measurement of the first hour postprandial distal antral motility index (MI), which is calculated as:
  MI = loge (sum of amplitude x number of contractions + 1) every 15 minutes following postcibal period (60 min).
  Effect size is the difference between means as a percentage of the mean index between the treatment groups. Estimated effect sizes are based on a paired t-test with the expected difference in mean of 1.6 motility index units in distal antral activity or 13.6% change in the antral motility index in ACTIVE compared to SHAM. It is to be noted that this is on a logarithmic scale and, therefore, a 10% change constitutes a clinically relevant difference.
  A higher MI value represents a better outcome.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: motility index units (see Description)
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
Number analyzed (Participants) | 6 | 6 | 6 | 6
motility index units (see Description) | 9.862 (1.549) | 10.38 (0.864) | 10.38 (1.469) | 8.433 (3.38)

2. Primary Outcome: Gastric Emptying of Solids - T1/2
Description: The median solid gastric emptying half-time in minutes from the stomach after a mixed meal as measured by scintigraphy.
  Approximately thirty minutes following ingestion of the Vibarnt / sham capsule, subjects ingested a standardized breakfast meal (320kcal egg, toast, milk) containing 99mTc. Anterior and posterior gamma camera images were obtained immediately following ingestion of the meal and every 15 minutes until 240 minutes.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
Number analyzed (Participants) | 6 | 6 | 6 | 5
Minutes | 120.7 (31.78) | 132.3 (34.38) | 134.7 (35.89) | 132.2 (43.91)

3. Secondary Outcome: Gastric Emptying at One Hour
Description: Gastric emptying scintigraphy (GES) is the 'gold standard' measurement for assessing stomach emptying rate.
  Stomach emptying was measured following ingestion of a standardized breakfast meal (320kcal egg, toast, milk) containing 99mTc.
  Anterior and posterior gamma camera images were obtained immediately following ingestion of the meal and every 15 minutes until 240 minutes.
  The outcome of GES at one hour is measuring the rate of solid emptying from the stomach after one hour in each of the study arms.
  A higher Fraction of solids emptying represents faster stomach emptying.
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: Fraction of solids emptying
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
Number analyzed (Participants) | 6 | 6 | 6 | 5
Fraction of solids emptying | 0.298 (0.0979) | 0.273 (0.0885) | 0.248 (0.0679) | 0.264 (0.0532)

4. Secondary Outcome: Gastric Emptying at Two Hours
Description: Gastric emptying scintigraphy (GES) is the 'gold standard' measurement for assessing stomach emptying rate.
  Stomach emptying was measured following ingestion of a standardized breakfast meal (320kcal egg, toast, milk) containing 99mTc.
  Anterior and posterior gamma camera images were obtained immediately following ingestion of the meal and every 15 minutes until 240 minutes.
  The outcome of GES at two hours is measuring the rate of solid emptying from the stomach after two hours in each of the study arms.
  A higher Fraction of solids emptying represents faster stomach emptying.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: Fraction of solids emptying
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
Number analyzed (Participants) | 6 | 6 | 6 | 4
Fraction of solids emptying | 0.495 (0.125) | 0.485 (0.168) | 0.457 (0.104) | 0.498 (0.177)

5. Secondary Outcome: Postprandial Distal Antral Motility Index
Description: First 0.5h postprandial distal antral motility index (Gastroduodenal Motility index (MI) MI formula: MI = loge (sum of amplitude x number of contractions + 1). Effect size is the difference between means as a percentage of the mean index between the treatment groups. Estimated effect sizes are based on a paired t-test with expected difference in mean of 1.6 motility index units in distal antral activity or 13.6% change in the antral motility index in ACTIVE compared to SHAM. It is to be noted that this is on a logarithmic scale and, therefore, an 10% change constitutes a clinically relevant difference.
  A higher MI value represents a better outcome.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: motility index units (See Description)
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
Number analyzed (Participants) | 6 | 6 | 6 | 6
motility index units (See Description) | 10.3 (1.102) | 10.38 (1.446) | 10.55 (1.532) | 10.34 (1.141)

ADVERSE EVENTS:
Time Frame: 6 hours
Arm/Group | Sham Vibrating Capsule | Vibrant Capsule (1 Vibration) | Vibrant Capsule (3 Vibration) | Vibrant Capsule (5 Vibration)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Permission to use study data is required

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT02736799/Prot_SAP_000.pdf